CLINICAL TRIAL: NCT06609551
Title: CtDNA-guided Selection of Adjuvant Chemotherapy Regimens for Elderly Colon Cancer Patients After Surgery: a Single-center, Randomized, Controlled Study
Acronym: ZJCH-CRCC-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhu Yuping, MD, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2024-380
Record Dates: First submitted 2024-09-22; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Colon Cancer; Colon Cancer (stage II & III)
Keywords: ctDNA (circulating tumor DNA); elderly colon cancer patients
MeSH Terms: conditions — Colonic Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm-A (No Intervention): Patients with negative ctDNA；Observation and follow-up
- Arm-B (Experimental): Patients with negative ctDNA;6-month adjuvant chemotherapy with 5-FU monotherapy
  Interventions: Drug: 6-month adjuvant chemotherapy with 5-FU monotherapy
- Arm-C (Experimental): Patients with positive ctDNA; 6-month adjuvant chemotherapy with 5-FU monotherapy
  Interventions: Drug: 6-month adjuvant chemotherapy with 5-FU monotherapy
- Arm-D (Experimental): Patients with positive ctDNA; XELOX intensive treatment group
  Interventions: Drug: XELOX intensive treatment group

INTERVENTIONS:
Drug: 6-month adjuvant chemotherapy with 5-FU monotherapy — 6 months of adjuvant chemotherapy with 5-FU monotherapy. The follow-up strategy for the four groups of subjects will be the same, including but not limited to chest plain or enhanced CT, abdominal/pelvic enhanced CT, and detection of the tumor marker carcinoembryonic antigen (CEA), until disease progression occurs. All patients will undergo peripheral blood ctDNA-MRD testing again six months after surgery.
  Arms: Arm-B; Arm-C
Drug: XELOX intensive treatment group — XELOX intensive treatment group. The follow-up strategy for the four groups of subjects will be the same, including but not limited to chest plain or enhanced CT, abdominal/pelvic enhanced CT, and detection of the tumor marker carcinoembryonic antigen (CEA), until disease progression occurs. All patients will undergo peripheral blood ctDNA-MRD testing again six months after surgery.
  Arms: Arm-D

SUMMARY:
The goal of this clinical trial is to explore the disease-free survival period of elderly patients with high-risk stage II and stage III colon cancer based on ctDNA detection. The main questions it aims to answer are:

Can ctDNA detection effectively guide the assessment of disease-free survival in elderly patients with high-risk stage II and stage III colon cancer? What is the correlation between postoperative ctDNA status and patient imaging as well as prognosis in elderly patients?

Secondary objectives include:

Evaluating the correlation between postoperative ctDNA status and patient imaging, as well as prognosis, in elderly patients.

Analyzing the positive rate of postoperative ctDNA and the ctDNA clearance rate.

Additionally, an exploratory objective of this study is to investigate recurrence models for postoperative patients.

Participants will undergo ctDNA testing to assess their disease status and will be monitored for disease-free survival. Imaging studies will also be conducted to correlate with ctDNA findings. The study aims to gain a deeper understanding of the role of ctDNA in predicting prognosis and monitoring disease recurrence in elderly patients with colon cancer.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial designed to explore the disease-free survival period of elderly patients with high-risk stage II and stage III colon cancer based on ctDNA detection.

1. Screening Phase Complete the routine pre-enrollment evaluation of subjects, such as medical history, pathological staging, and treatment history. Researchers will assess whether subjects meet the enrollment criteria (see inclusion and exclusion criteria). For subjects who meet the enrollment criteria, the attending physician will inform the subjects and their families, explaining the purpose, advantages, disadvantages, and the entire research process of this clinical trial. They will seek the opinions of the subjects and their families, and obtain signed informed consent from the subjects.

   Researchers need to collect baseline postoperative tissue samples for detection, which will be used for the customization of personalized probes for subsequent blood tests.
2. Adjuvant Therapy/Follow-up Phase Elderly colorectal cancer patients who meet the inclusion and exclusion criteria will undergo ctDNA-MRD testing after surgery. ctDNA-negative patients will be randomly divided into two groups in a 1:1 ratio: 1) Observation and follow-up; 2) 6-month adjuvant chemotherapy with 5-FU monotherapy. Patients who test positive for ctDNA will be randomly assigned in a 1:1 ratio to receive: 1) 6 months of 5-FU monotherapy; 2) XELOX intensive treatment group. The follow-up strategy is the same for all four groups, including but not limited to chest plain or enhanced CT, abdominal/pelvic enhanced CT, and detection of the tumor marker carcinoembryonic antigen (CEA) until disease progression occurs. All patients will undergo peripheral blood ctDNA-MRD testing again half a year after surgery.
3. Management Measures for Subjects with Disease Progression If a patient experiences disease progression, efforts should be made to continue tracking and recording the patient's subsequent anti-tumor treatment and survival outcomes, including local and/or systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 70-80, both male and female are eligible;
2. Patients with histopathologically confirmed stage II high-risk or stage III colon cancer;
3. Patients with an ECOG score of ≤2;
4. Patients who are required to undergo tissue genetic testing;
5. Subjects who voluntarily participate in this study, sign the informed consent form, have good compliance, and cooperate with follow-up visits.

Exclusion Criteria:

1. Patients with one or more severe concomitant systemic diseases that, in the investigator's opinion, would impair the patient's ability to complete the study.
2. Patients who have had a history of malignant tumors within 5 years.
3. Any unstable systemic disease (including active infection, poorly controlled diabetes, poorly controlled hypertension, unstable angina, congestive heart failure, myocardial infarction within one year, severe arrhythmia requiring medical treatment, liver, kidney, or metabolic diseases).
4. Patients suffering from severe mental illnesses.
5. Patients who have participated in other clinical trials within 30 days prior to screening.
6. Patients who are unable to undergo adjuvant chemotherapy.

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 312 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year DFS (Disease-Free Survival) | From enrollment to the end of treatment at 2 years
  Disease-free survival (DFS): the time from the start of treatment to the progression of the disease.

SECONDARY OUTCOMES:
5-year DFS (Disease-Free Survival) | From enrollment to the end of treatment at 5 years
  Disease-free survival (DFS): the time from the start of treatment to the progression of the disease.
2-year OS (Overall Survival) | From enrollment to the end of treatment at 2 years
  Overall Survival (OS) refers to the total survival time from the start of treatment until death directly caused by the disease.
5-year OS (Overall Survival) | From enrollment to the end of treatment at 5 years
  Overall Survival (OS) refers to the total survival time from the start of treatment until death directly caused by the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Badia-Ramentol J, Linares J, Gomez-Llonin A, Calon A. Minimal Residual Disease, Metastasis and Immunity. Biomolecules. 2021 Jan 20;11(2):130. doi: 10.3390/biom11020130. PMID 33498251
- [Background] Dasari A, Morris VK, Allegra CJ, Atreya C, Benson AB 3rd, Boland P, Chung K, Copur MS, Corcoran RB, Deming DA, Dwyer A, Diehn M, Eng C, George TJ, Gollub MJ, Goodwin RA, Hamilton SR, Hechtman JF, Hochster H, Hong TS, Innocenti F, Iqbal A, Jacobs SA, Kennecke HF, Lee JJ, Lieu CH, Lenz HJ, Lindwasser OW, Montagut C, Odisio B, Ou FS, Porter L, Raghav K, Schrag D, Scott AJ, Shi Q, Strickler JH, Venook A, Yaeger R, Yothers G, You YN, Zell JA, Kopetz S. ctDNA applications and integration in colorectal cancer: an NCI Colon and Rectal-Anal Task Forces whitepaper. Nat Rev Clin Oncol. 2020 Dec;17(12):757-770. doi: 10.1038/s41571-020-0392-0. Epub 2020 Jul 6. PMID 32632268
- [Background] Ueda Y, Shiraishi N, Kawasaki T, Akagi T, Ninomiya S, Shiroshita H, Etoh T, Inomata M. Short- and long-term outcomes of laparoscopic surgery for colorectal cancer in the elderly aged over 80 years old versus non-elderly: a retrospective cohort study. BMC Geriatr. 2020 Nov 4;20(1):445. doi: 10.1186/s12877-020-01779-2. PMID 33148215
- [Background] Argiles G, Tabernero J, Labianca R, Hochhauser D, Salazar R, Iveson T, Laurent-Puig P, Quirke P, Yoshino T, Taieb J, Martinelli E, Arnold D; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Localised colon cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2020 Oct;31(10):1291-1305. doi: 10.1016/j.annonc.2020.06.022. Epub 2020 Jul 20. No abstract available. PMID 32702383
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Hutchins LF, Unger JM, Crowley JJ, Coltman CA Jr, Albain KS. Underrepresentation of patients 65 years of age or older in cancer-treatment trials. N Engl J Med. 1999 Dec 30;341(27):2061-7. doi: 10.1056/NEJM199912303412706. PMID 10615079
- [Background] Kim JH. Chemotherapy for colorectal cancer in the elderly. World J Gastroenterol. 2015 May 7;21(17):5158-66. doi: 10.3748/wjg.v21.i17.5158. PMID 25954089
- [Background] Herrera AP, Snipes SA, King DW, Torres-Vigil I, Goldberg DS, Weinberg AD. Disparate inclusion of older adults in clinical trials: priorities and opportunities for policy and practice change. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S105-12. doi: 10.2105/AJPH.2009.162982. Epub 2010 Feb 10. PMID 20147682
- [Background] Waldron RP, Donovan IA, Drumm J, Mottram SN, Tedman S. Emergency presentation and mortality from colorectal cancer in the elderly. Br J Surg. 1986 Mar;73(3):214-6. doi: 10.1002/bjs.1800730320. PMID 3947921
- [Background] Dekker JW, van den Broek CB, Bastiaannet E, van de Geest LG, Tollenaar RA, Liefers GJ. Importance of the first postoperative year in the prognosis of elderly colorectal cancer patients. Ann Surg Oncol. 2011 Jun;18(6):1533-9. doi: 10.1245/s10434-011-1671-x. Epub 2011 Mar 29. PMID 21445672
- [Background] Zheng R, Zhang S, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2016. J Natl Cancer Cent. 2022 Feb 27;2(1):1-9. doi: 10.1016/j.jncc.2022.02.002. eCollection 2022 Mar. PMID 39035212
- [Background] Kurniali PC, Hrinczenko B, Al-Janadi A. Management of locally advanced and metastatic colon cancer in elderly patients. World J Gastroenterol. 2014 Feb 28;20(8):1910-22. doi: 10.3748/wjg.v20.i8.1910. PMID 24616568
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338